CLINICAL TRIAL: NCT00722488
Title: An Open-Label, Dose Escalation, Phase I Study of MLN4924, a Novel Inhibitor of Nedd8 Activating Enzyme, in Adult Patients With Lymphoma or Multiple Myeloma
Brief Title: Study of MLN4924, a Novel Inhibitor of Nedd8 Activating Enzyme, in Adult Patients With Lymphoma or Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C15002
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Hematologic Malignancies; Multiple Myeloma; Lymphoma; Hodgkin Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Multiple Myeloma; Lymphoma; Hodgkin Disease | interventions — pevonedistat

ARMS (1):
- 1 (Experimental): MLN4924
  Interventions: Drug: MLN4924

INTERVENTIONS:
Drug: MLN4924 — Intravenous dose 100 mg/m2 on a Days 1,4,8,11 schedule within a 21-day treatment cycle. Treatment may continue until disease progression or unacceptable toxicity develops.

SUMMARY:
This is an open-label, multicenter, phase 1, dose escalation study of MLN4924 in adult patients with lymphoma or multiple myeloma. The patient population will consist of adults with a confirmed diagnosis of lymphoma (Waldenstrom's macroglobulinemia is permitted) or multiple myeloma that is relapsed and/or refractory after at least 2 prior standard chemotherapeutic regimens and for which no curative option exists.

Patients in the expansion cohort, Schedule E, must specifically have Hodgkin lymphoma, DLBCL-GCB subtype, DLBCL-non-GCB subtype, or Mantle Cell Lymphoma (MCL). Patients with multiple myeloma will no longer be evaluated as a part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Patients must have a confirmed diagnosis of lymphoma (Waldenstrom's macroglobulinemia is permitted) or multiple myeloma that is relapsed and/or refractory after at least 2 prior standard chemotherapeutic regimens and for which no curative option exists.

  1. As of Protocol Amendment 7, patients in the expansion cohort, Schedule E, must specifically have Hodgkin lymphoma, DLBCL-GCB subtype, DLBCL-non-GCB subtype, or Mantle Cell Lymphoma (MCL). Patients with multiple myeloma will no longer be evaluated as a part of this study.
* Tumor that is evaluable by radiography, serum or urine electrophoresis (for patients with multiple myeloma), or clinical evaluations.

  1. As of Protocol Amendment 7, tumor that is evaluable by radiography or clinical evaluations.
* Suitable venous access for the conduct of blood sampling for MLN4924
* Adequate Organ Function

Exclusion Criteria:

* Systemic antineoplastic therapy within 21 days preceding first dose of study treatment, or rituximab therapy within 2 months preceding first dose of study treatment (unless there was evidence of PD since their last dose of rituximab).
* Treatment with corticosteroids within 7 days preceding first dose of study treatment.
* Prior treatment with radiation therapy involving >25% of bone marrow; Any radiotherapy within 14 days before first dose of study treatment.
* Treatment with CYP3A inducers within 14 days before the first dose of MLN4924. Moderate and strong CYP3A inhibitors and CYP3A inducers are not permitted during the study.
* Patients requiring Coumadin who cannot be switched to a low molecular weight heparin should not be considered for this study.
* Absolute neutrophil count less than 1,000/mm3; platelet count less than 75,000/mm3.
* Calculated creatinine clearance less than or equal to 50 mL/minute.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-06; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and tolerability | 12 months (maximum duration of therapy)

SECONDARY OUTCOMES:
Disease response | 12 months (maximum duration of therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Winship Cancer Institute, Atlanta, Georgia
  - Roswell Park Cancer Institute, Buffalo, New York

REFERENCES:
- [Derived] Faessel HM, Mould DR, Zhou X, Faller DV, Sedarati F, Venkatakrishnan K. Population pharmacokinetics of pevonedistat alone or in combination with standard of care in patients with solid tumours or haematological malignancies. Br J Clin Pharmacol. 2019 Nov;85(11):2568-2579. doi: 10.1111/bcp.14078. Epub 2019 Sep 4. PMID 31355467